CLINICAL TRIAL: NCT05769816
Title: A Novel Combination Therapeutic Strategy Aiming to Functional Cure for Chronic Hepatitis B Virus Infection (Sustained HBsAg Loss) (A)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: The Affiliated Hospital Of Southwest Medical University (Other); Guizhou Provincial People's Hospital (Other); Chongqing Three Gorges Central Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0220
Record Dates: First submitted 2023-02-22; First posted 2023-03-15 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Chronic Hepatitis b; Anti-PD-1 Antibody
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — spartalizumab; nas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): NAs combined with anti-PD-1 antibody, followed by NAs monotherapy
  Interventions: Drug: Anti-PD-1 antibody; Drug: NAs
- Group 2 (Active Comparator): NAs
  Interventions: Drug: NAs

INTERVENTIONS:
Drug: Anti-PD-1 antibody — Once/two or three weeks, dose lower than the dose used in cancer patients, subcutaneous/intravenous injection
  Arms: Group 1
Drug: NAs — Once/day, 1 capsule/time, oral
  Other Names: ETV/TDF/TAF

SUMMARY:
Hepatitis B virus (HBV) infection is a major public health threat in China. At present, a functional cure, also known as clinical cure or sustained Hepatitis B surface antigen (HBsAg) loss, is recommended as the ideal endpoint of HBV treatment. However, HBsAg loss can be achieved in less than 10% of chronic hepatitis B (CHB) patients treated with current available antiviral drug interferon (IFNα) or nucleos(t)ide analogues (NAs) monotherapy. With the support of the national major special funding for infectious diseases from "11th Five-Year Plan" to "13th Five-Year Plan", we have implemented a pioneer clinical study of sequential combination of IFNα therapy on NAs to treat NAs-treated CHB patients (ie. New Switch Study). This is the world's first clinical trial aiming to functional cure, which increased the rate of HBsAg loss to 15% in the overall population in our study, and to 30-50% among those with lower baseline HBsAg levels. How to further improve the HBsAg loss rate is an urgent issue for us. The key point of achieving functional cure is to reverse the HBV-specific T cell exhaustion and establish the long-term immune control against HBV infection. Programmed death-1 (PD-1)/ programmed death-ligand 1 (PD-L1) axis blockade has been demonstrated to reinvigorate exhausted CD8+ T cells, and would be a potential strategy to treat chronic HBV infection. In this study, a large multicenter prospective study will be performed to explore the safety and efficacy of a novel combination strategy involving immune checkpoint inhibitor (anti-PD-1 antibody) in CHB patients, observe the HBsAg loss rate in NA-treated CHB patients receiving this combination strategy, evaluate the potential of breaking immune tolerance by this strategy, and further assess its efficacy to further improve the clinical cure rate on the basis of New Switch Study. Based on New Switch Study, this study further attempts to reverse T cell exhaustion in CHB patients, explore a novel platform of combination therapy development for clinical cure, and ultimately increase the HBsAg loss rate to higher than 50% in overall patients. The implementation of the project is expected to reduce the burden of HBV infection in China and contribute to the goal of global elimination of hepatitis B and C by 2030 (WHO 2030).

ELIGIBILITY:
Inclusion Criteria:

* 1) Sign the informed consent form before inclusion and be able to complete the study according to the study requirements;
* 2) From inclusion to 30 days after the last administration of the study drug, male subjects or female subjects of childbearing age are willing to voluntarily take effective contraceptive measures;
* 3) 18-70 years old. The weight of male subjects is not less than 45 kg, and the weight of female subjects is not less than 40 kg. Body mass index (BMI) is within the range of 18-32 kg/m^2;
* 4) NAs-naive/NAs-experienced CHB patients.

Exclusion Criteria:

* 1) A history of allergy, or who are suspected by the researcher to be allergic to the active ingredient of the drug under study or its excipients;
* 2) Use of inhibitors, inducers or substrates of CYP3A4 within 28 days before enrollment;
* 3) Systematical use of immunosuppressants, immunomodulators (thymosin) and cytotoxic drugs within 6 months before enrollment, or vaccination of live attenuated vaccine within 1 month before enrollment;
* 4) Acute infection within 2 weeks before enrollment which requires intravenous antibiotic treatment, or existing infection which requires anti-infection treatment when enrollment;
* 5) Clinically significant acute and chronic liver disease not caused by HBV infection (judged by reseachers);
* 6) Confirmed or suspected decompensated cirrhosis, including but not limited to: hepatic encephalopathy, hepatorenal syndrome, bleeding from esophageal varices, splenomegaly, ascites, etc, or evidence of progressive liver fibrosis;
* 7) Primary liver cancer, or alpha-fetoprotein (AFP) is greater than 50 ug/L or imaging suggests the possibility of malignant liver lesions, or other malignant tumors or a history of other malignant tumors within 5 years before enrollment (except that the malignant tumors have been completely relieved after treatment and patients have not received additional medical or surgical intervention within 3 years before screening);
* 8) A history of pathological fracture or osteoporosis;
* 9) Gastrointestinal dysfunction or gastrointestinal diseases that might affect the absorption of oral drugs, such as severe gastric ulcer, erosive gastritis, partial gastrectomy, and persistent gastrointestinal symptoms (such as nausea, vomiting, or diarrhea) >2 grades;
* 10) Serious diseases of circulatory, respiratory, urinary, blood, metabolic, immune, mental, neurological, renal and other systems;
* 11) Major trauma or major surgery within 3 months before enrollment, or planned surgery during the study period;
* 12) Blood donation/loss ≥ 400 mL within 3 months before enrollment, or given a blood transfusion within 3 months before enrollment, or blood donation/loss ≥ 200 mL within 1 month before enrollment;
* 13) Platelet count<90 × 10^9/L, white blood cell count<3.0 × 10^9/L, neutrophil count<1.3 × 10^9/L, total serum bilirubin>2 × upper limit of normal (ULN), albumin<30 g/L, creatinine clearance ≤ 60 mL/min (calculated by CKD-EPI formula), or international normalized ratio of prothrombin time (INR)>1.5 (unless receiving stable anticoagulant therapy);
* 14) Hepatitis C virus (HCV) antibody (+), HIV antigen/antibody (+), or treponema pallidum antibody (+) and rapid plasma regain (RPR) test (+);
* 15) A history of continuous alcohol abuse within 3 years before enrollment (average daily alcohol consumption exceeds 20 gram);
* 16) A history of drug dependence or drug abuse within 1 year before enrollment;
* 17) Those who have participated in clinical trials of other investigational drugs or medical devices and taken investigational drugs or used medical devices within 3 months before enrollment;
* 18) Female in suckling period or pregnancy test (+) during screening;
* 19) Subjects who are considered by the researcher to have other factors that are not suitable for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum HBsAg | Baseline
  Serum HBsAg level
Serum HBsAg | 24 weeks after the treatment
  Serum HBsAg level
Serum HBsAg | 48 weeks after the treatment
  Serum HBsAg level
Serum HBsAg | 24 weeks after the end of treatment
  Serum HBsAg level
Serum HBV DNA | Baseline
  Serum HBV DNA level
Serum HBV DNA | 24 weeks after the treatment
  Serum HBV DNA level
Serum HBV DNA | 48 weeks after the treatment
  Serum HBV DNA level
Serum HBV DNA | 24 weeks after the end of treatment
  Serum HBV DNA level
Serum alanine aminotransferase (ALT) | Baseline
  Serum ALT level
Serum alanine aminotransferase (ALT) | 24 weeks after the treatment
  Serum ALT level
Serum alanine aminotransferase (ALT) | 48 weeks after the treatment
  Serum ALT level
Serum alanine aminotransferase (ALT) | 24 weeks after the end of treatment
  Serum ALT level

OTHER OUTCOMES:
Other HBV markers | Baseline
  Levels of other HBV markers
Other HBV markers | 24 weeks after the treatment
  Levels of other HBV markers
Other HBV markers | 48 weeks after the treatment
  Levels of other HBV markers
Other HBV markers | 24 weeks after the end of treatment
  Levels of other HBV markers
Immune response of T and B cells | Baseline
  Frequencies and functions of T and B cells (tested by flowcytometry/FluoroSpot/ELISPOT)
Immune response of T and B cells | 24 weeks after the treatment
  Frequencies and functions of T and B cells (tested by flowcytometry/FluoroSpot/ELISPOT)
Immune response of T and B cells | 48 weeks after the treatment
  Frequencies and functions of T and B cells (tested by flowcytometry/FluoroSpot/ELISPOT)
Immune response of T and B cells | 24 weeks after the end of treatment
  Frequencies and functions of T and B cells (tested by flowcytometry/FluoroSpot/ELISPOT)
Virus and host genome | Baseline
  Detect virus and host genome (focusing on HBV genotype, resistant mutation) using peripheral blood by sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ren, MM, Study Director — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The 2nd affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He T, Chen M, Liu M, Zhang L, Sun H, Zhang L, Li A, Zeng W, Ling N, Shi X, He H, Peng M, Cai D, Hu P, Zhang D, Lan Y, Ren H. Twenty-four-week anti-PD-1 antibody regimen promoted HBsAg reduction and concurrently enhanced HBV-specific T cell responses in patients with chronic hepatitis B. Gut. 2025 Dec 24:gutjnl-2025-336655. doi: 10.1136/gutjnl-2025-336655. Online ahead of print. PMID 41443982